CLINICAL TRIAL: NCT05716412
Title: Personality and Vulnerability for Affective Spectrum Disorders and Complaints: The Role of Gene-Environment Correlations (rGE) and Interactions (GxE)
Brief Title: Gene-environment Interactions in Families With Adolescents (Gen-omgevingsinteracties in Gezinnen Met Adolescenten)
Acronym: GiGA
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Fund for Scientific Research, Flanders, Belgium (Other)
Responsible Party: Sponsor
Other Study IDs: S56106
Record Dates: First submitted 2014-05-19; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2016-05

CONDITIONS: Affective Spectrum Symptoms

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Saliva

GROUPS / COHORTS (3):
- Adopted adolescents and their adoptive parents: Adopted before the age of one, currently between 12 to 18 years old
- Adolescents and their biological related parents: Matched to adoptive adolescents
- Additional community sample

SUMMARY:
English:

The main purpose of this study is to investigate the developmental trajectories of parents and adolescents in the Flemish region of Belgium. The investigators will focus on the role of genetic factors, environmental factors (e.g. parental rearing styles), and the interaction between these factors. Specifically, it will be investigated were difficulties or strengths in the development of adolescents can be attributed to. How an individual's genetic characteristics and his/her family environment can interact, will also be monitored. This study is closely related to the Leuvense Adoption Study (http://leuvenseadoptiestudie.be/). Just like this research, the investigators will take child and parent factors in account, as well as their interaction. The investigators will not only focus on vulnerability, but also on protective factors that can give resilience to both parents and children. The theoretical framework of this study is twofold. (1) In the development of children, genes and environment are interwoven in a dynamical relation. Neither genes or environment alone can explain how a child will develop over time. (2) The relation between genetic and environmental factors can be expressed in different ways. On the one hand, a certain genetic contribution can impact the way parents will uphold a certain parental rearing style. On the other hand, having certain genetic characteristics will have consequences for how adolescents will react to their environment. For example, a certain parental rearing style will strengthen some adolescents resilience, but for other adolescents this could equally lead to a more maladaptive development. Thus, depending on his or her genetic endowment, a child will develop differently given a certain family environment.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents adopted before the age of one and currently 12 to 18 years old (from international adoption) and their adoptive parents
* Matched community sample of adolescents between the age of 12 and 18 years old and their biological related parents

Exclusion Criteria:

* Major medical or psychiatric disease

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adopted adolescents and their parents, adolescents with their biological parents, and an additional community sample.
Sampling Method: Non-Probability Sample
Enrollment: 1326 (Actual)
Dates: Start 2014-09; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Beck's Depression Inventory / Children's Depression Inventory | current symptoms, measured once after enrollment
  Dimensional assessment and cut-off scores using Beck's Depression Inventory for the adults and Kovacs' Children's Depression Inventory for the adolescents.

SECONDARY OUTCOMES:
Somatic Symptoms Questionnaire | current complaints, measured once after enrollment
  Pain and fatigue related complaints. Sometimes referred to as somatic complaints.
Depressive Experiences Questionnaire: self-criticism and dependency | measured once after enrollment
  Personality assessment by Blatt's polarities of experience model. Blatt's model is a two-polarity model: relatedness (dependency) and self-definition (self-criticism).

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Luyten, Prof. Dr., Principal Investigator — KU Leuven - Faculty of Psychology and Educational Sciences - Clinical Psychology Research Unit
Locations (2):
- Belgium (2):
  - University of Gent - Faculty of Psychology and Educational Sciences - Department of Developmental-, Personality- and Social Psychology, Ghent, Oost-Vlaanderen
  - KU Leuven - Department of Psychology and Educational Sciences - Clinical Psychology Research Unit, Leuven, Vlaams-Brabant